CLINICAL TRIAL: NCT01291849
Title: The Effect-site Concentration of Remifentanil for Preventing Cough During Emergence From Balanced Anesthesia for Nasal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Wyun-Kon Park/Professor, Yonsei University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2009-0578
Record Dates: First submitted 2011-02-01; First posted 2011-02-09 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-01

CONDITIONS: Cough
Keywords: nasal surgery; endoscopic sinus surgery; septoplasty; Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- remifentanil for intranasal surgery (Experimental)
  Interventions: Drug: Dixon up-and-down method

INTERVENTIONS:
Drug: Dixon up-and-down method — The target Ce of remifentanil was determined by the response of the previous patient using Dixon's up-and-down method. If the patients did not cough throughout peri-extubation period, the extubation was defined as a smooth emergence, and the predetermined concentration of remifentanil for the subsequent patient was decreased by 0.5 ng ml-1. Similarly, if the patient cough anytime around extubation it was considered as failed smooth emergence and the predetermined concentration was increased by 0.5 ng ml-1 for the next patient. The patients were enrolled until getting at least six cross-over pairs in Dixon sequential allocation method.

SUMMARY:
After nasal surgery, emergence cough or straining will produce venous engorgement and increase bleeding from the surgical site, so the necessity for smooth extubation without severe cough during emergence provides a challenge for the anesthetists. Recently, remifentanil is commonly used short-acting opioid, and several studies have demonstrated the antitussive effect of remifentanil via effect-site target-controlled infusion during emergence. However, there may be gender difference in response to opioid, and the previous studies about antitussive effect of remifentanil are targeted at female patients and there is no investigation of effect site concentration of remifentanil for male patients undergoing nasal surgery. The purpose of this study is to evaluate the effect-site concentration of remifentanil via target-controlled infusion for preventing cough in man after sevofluorane balanced anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* all male aged 18-60 years
* ASA(American Society of Anesthesiologists)physical status I or II
* who underwent ESS(endoscopic sinus surgery)or septoplasty under sevoflurane-remifentanil balanced anesthesia

Exclusion Criteria:

* predicted difficult airway,
* BMI(Body Mass Index) of more than 30 kg/m2,
* chronic respiratory disease,
* recent respiratory track infection,
* chronic coughing,
* significant cardiovascular,
* hepatic or renal disease,
* current smokers
* medical history of medication of opioid or ACEI(angiotensin covering enzyme inhibitor)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
cough incidence | from sevoflurane discontinuation (at the end of anesthesia) to 5 min after extubation
  Cough is defined as a strong and sudden contraction of the abdomen or forced exhalation movement.
cough grade | from sevoflurane discontinuation (at the end of anesthesia) to 5 min after extubation
  Cough occurrence and number are recorded according to the grading system as follow; Grade 0 - no cough Grade 1 - light (single) cough Grade 2 - moderate cough (more than 1 episode of non-sustained cough) Grade 3 - sustained and repetitive cough movement and head lift.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Lee B, Lee JR, Na S. Targeting smooth emergence: the effect site concentration of remifentanil for preventing cough during emergence during propofol-remifentanil anaesthesia for thyroid surgery. Br J Anaesth. 2009 Jun;102(6):775-8. doi: 10.1093/bja/aep090. Epub 2009 May 2. PMID 19411668